CLINICAL TRIAL: NCT02513550
Title: A Multicenter, Randomized, Double-Blind Study Comparing the Efficacy and Safety of Ixekizumab Dosing Regimens in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study Comparing Different Dosing Regimens of Ixekizumab (LY2439821) in Participants With Moderate to Severe Plaque Psoriasis
Acronym: IXORA-P
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15988; I1F-MC-RHBP (Other: Eli Lilly and Company); 2015-000190-12 (EudraCT Number)
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 80 mg Ixekizumab Q2W (Experimental): 160 milligrams (mg) ixekizumab given as 2 subcutaneous (SQ) injections at baseline and then 80 mg ixekizumab given as 1 SQ injection every 2 weeks (Q2W) to week 52. Placebo administered SQ, Q2W to maintain blind.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- 80 mg Ixekizumab Q4W (Experimental): 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection every 4 weeks (Q4W) to week 52. Placebo administered SQ, Q2W to maintain blind.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- 80 mg Ixekizumab Q4W/Q2W (Experimental): 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as one SQ injection Q4W with step-up dosing to Q2W as needed (Q4W/Q2W step-up) to week 52. Placebo administered SQ, Q2W to maintain blind.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- 80 mg Ixekizumab Q2W Maximum Extended Enrollment (ME2) Cohort (Experimental): 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q2W to week 52. Placebo administered SQ, Q2W to maintain blind.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- 80 mg Ixekizumab Q4W Maximum Extended Enrollment Cohort (Experimental): 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q4W to week 52. Placebo administered SQ, Q2W to maintain blind.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- 80 mg Ixekizumab Q4W/Q2W Maximum Extended Enrollment Cohort (Experimental): 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as one SQ injection Q4W with step-up dosing to Q2W as needed (Q4W/Q2W step-up) to week 52. Placebo administered SQ, Q2W to maintain blind.
  Interventions: Drug: Ixekizumab; Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SQ
  Other Names: LY2439821
Drug: Placebo — Administered SQ

SUMMARY:
The main purpose of this study is to evaluate the efficacy of ixekizumab dosing regimens in participants with plaque psoriasis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate both the safety and efficacy of ixekizumab dosing regimens. There are 3 study periods: Screening Period, Blinded Treatment Dosing Period, and Post-Treatment Follow-Up.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque psoriasis for at least 6 months prior to enrollment
* At least 10% BSA of psoriasis at screening and at enrollment
* sPGA score of at least 3 and PASI score of at least 12 at screening and at enrollment
* Candidates for phototherapy and/or systemic therapy
* Participant must agree to use reliable method of birth control during the study; women must continue using birth control for at least 12 weeks after stopping treatment

Exclusion Criteria:

* Predominant pattern of pustular, erythrodermic, or guttate forms of psoriasis
* History of drug-induced psoriasis
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to enrollment and during the study
* Received systemic non-biologic psoriasis therapy or phototherapy within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks prior to enrollment
* Concurrent or recent use of any biologic agent
* Have participated in any study with ixekizumab
* Received a live vaccination within 12 weeks prior to enrollment
* Serious disorder or illness other than psoriasis
* Ongoing or serious infection within the last 12 weeks or evidence of tuberculosis
* Major surgery within 8 weeks of baseline, or will require surgery during the study
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (124):
- United States (58):
  - Total Skin and Beauty Dermatology Center PC, Birmingham, Alabama
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - David Stoll, M.D., Beverly Hills, California
  - Dermatology Research Associates, Los Angeles, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Cherry Creek Research, Inc, Denver, Colorado
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Avail Clinical Research LLC, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - University of South Florida, Tampa, Florida
  - Advanced Medical Research, Atlanta, Georgia
  - University Dermatology, Darien, Illinois
  - Deaconess Clinic Inc, Evansville, Indiana
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Dermatology Specialist, Louisville, Kentucky
  - Dr. Shondra Smith MD, Lake Charles, Louisiana
  - DermAssociates, P.C., Rockville, Maryland
  - ActivMed Practices & Research, Inc, Beverly, Massachusetts
  - Central Dermatology PC, St Louis, Missouri
  - ActivMed Practices & Research, Inc, Newington, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Mount Sinai School of Medicine Dermatology Clinical Trials, New York, New York
  - Skin Search of Rochester, Inc, Rochester, New York
  - University of North Carolina Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Healthcare Research Consultant, Tulsa, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pennsylvania Regional Center for Arthritis & Osteoarthritis, Wyomissing, Pennsylvania
  - Yardley Dermatology, Yardley, Pennsylvania
  - Clinical Partners LLC, Johnston, Rhode Island
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - The Skin Wellness Center PC, Knoxville, Tennessee
  - Austin Dermatology Associates, Austin, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Pflugerville Dermatology Clinical Research Center, Pflugerville, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - Virginia Clinical Research, Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
  - Multicare Health System, Tacoma, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
- Australia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Benowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carlton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darlinghurst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fremantle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phillip
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloongabba
- Canada (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Markham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oakville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peterborough
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond Hill
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Windsor
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nový Jičín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plzen-Bory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darmstadt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mahlow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orosháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szolnok
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takaoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tsu
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morelia
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kielce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Świdnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (5):
  - Office of Dr. Samuel Sanchez PSC, Caguas
  - Office of Dr. Alma M. Cruz, Carolina
  - Ponce School of Medicine CAIMED Center, Ponce
  - GCM Medical Group PSC, San Juan
  - Mindful Medical Research, San Juan
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Constanța
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Click here for more information about this study: A Study Comparing Different Dosing Regimens of Ixekizumab (LY2439821) in Participants With Moderate to Severe Plaque Psoriasis — http://www.lillytrialguide.com/EN-us/studies/psoriasis/rhbp

RESULTS

PARTICIPANT FLOW:
Groups:
- 80 mg Ixekizumab Q4W: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q4W to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q2W; 80 mg Ixekizumab Q2W Maximum Extended Enrollment Cohort: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q2W to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q4W Maximum Extended Enrollment Cohort: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80mg ixekizumab given as 1 SQ injection Q4W to week 52. Placebo administered SQ, Q2W to maintain blind.
Period: Double Blind Treatment Period
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W | 80 mg Ixekizumab Q4W Maximum Extended Enrollment Cohort | 80 mg Ixekizumab Q4W/Q2W Maximum Extended Enrollment Cohort | 80 mg Ixekizumab Q2W Maximum Extended Enrollment Cohort
Started | 310 | 306 | 611 | 9 | 5 | 16
Received at Least One Dose of Study Drug | 310 | 306 | 609 | 9 | 5 | 16
Completed | 274 | 268 | 537 | 9 | 4 | 15
Not Completed | 36 | 38 | 74 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 11 | 11 | 25 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 13 | 17 | 0 | 1 | 0
Not completed — Lost to Follow-up | 9 | 7 | 11 | 0 | 0 | 1
Not completed — Lack of Efficacy | 4 | 5 | 6 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 4 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 4 | 0 | 0 | 0
Not completed — Site terminated by sponsor | 1 | 1 | 3 | 0 | 0 | 0
Not completed — Met exclusion criteria and was not dosed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Due to personal business | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 2 | 0 | 0 | 0
Period: Post-Treatment Follow-up Period
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W | 80 mg Ixekizumab Q4W Maximum Extended Enrollment Cohort | 80 mg Ixekizumab Q4W/Q2W Maximum Extended Enrollment Cohort | 80 mg Ixekizumab Q2W Maximum Extended Enrollment Cohort
Started | 285 (Participants who discontinued double blind phase had an option to enter post-treatment phase.) | 283 (Participants who discontinued double blind phase had an option to enter post-treatment phase.) | 559 (Participants who discontinued double blind phase had an option to enter post-treatment phase.) | 9 (Participants who discontinued double blind phase had an option to enter post-treatment phase.) | 4 (Participants who discontinued double blind phase had an option to enter post-treatment phase.) | 15 (Participants who discontinued double blind phase had an option to enter post-treatment phase.)
Completed | 254 | 244 | 496 | 9 | 4 | 15
Not Completed | 31 | 39 | 63 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 20 | 26 | 0 | 0 | 0
Not completed — Early terminated but completed follow-up | 12 | 16 | 20 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 2 | 7 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 4 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Subject move out of town | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Subject did not come for Visit-802 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Labor Reasons | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W | 80 mg Ixekizumab Q4W Maximum Extended Enrollment Cohort | 80 mg Ixekizumab Q4W/Q2W Maximum Extended Enrollment Cohort | 80 mg Ixekizumab Q2W Maximum Extended Enrollment Cohort | Total
Number analyzed (Participants) | 310 | 306 | 611 | 9 | 5 | 16 | 1257
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All randomized participants who received at least one dose of study drug and had baseline age data.
  years
    number analyzed (Participants) | 310 | 306 | 609 | 9 | 5 | 16 | 1255
    (all) | 47.4 (13.50) | 45.9 (12.85) | 49.0 (13.61) | 40.0 (9.62) | 46.0 (13.17) | 46.1 (13.05) | 47.8 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 107 | 199 | 2 | 0 | 4 | 423
  Male | 199 | 199 | 412 | 7 | 5 | 12 | 834
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 55 | 111 | 0 | 0 | 0 | 225
  Not Hispanic or Latino | 243 | 244 | 489 | 9 | 5 | 16 | 1006
  Unknown or Not Reported | 8 | 7 | 11 | 0 | 0 | 0 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 12 | 23 | 0 | 0 | 0 | 46
  Asian | 31 | 32 | 64 | 9 | 5 | 16 | 157
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 4 | 0 | 0 | 0 | 4
  Black or African American | 14 | 8 | 22 | 0 | 0 | 0 | 44
  White | 251 | 253 | 486 | 0 | 0 | 0 | 990
  More than one race | 3 | 1 | 12 | 0 | 0 | 0 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 14 | 16 | 29 | 0 | 0 | 0 | 59
  Argentina | 9 | 9 | 19 | 0 | 0 | 0 | 37
  Romania | 5 | 5 | 9 | 0 | 0 | 0 | 19
  Hungary | 11 | 10 | 23 | 0 | 0 | 0 | 44
  United States | 119 | 118 | 238 | 0 | 0 | 0 | 475
  Czechia | 3 | 3 | 8 | 0 | 0 | 0 | 14
  Japan | 5 | 2 | 9 | 0 | 0 | 0 | 16
  Canada | 49 | 49 | 99 | 0 | 0 | 0 | 197
  South Korea | 11 | 12 | 22 | 9 | 5 | 16 | 75
  Taiwan | 5 | 6 | 9 | 0 | 0 | 0 | 20
  Poland | 43 | 43 | 83 | 0 | 0 | 0 | 169
  Mexico | 10 | 8 | 17 | 0 | 0 | 0 | 35
  Australia | 14 | 14 | 28 | 0 | 0 | 0 | 56
  Germany | 12 | 11 | 18 | 0 | 0 | 0 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) of (0,1)
Description: The sPGA is the physician's determination of the participant's Psoriasis (Ps) lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's Ps was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline. Participants who did not meet the clinical response criteria or had missing data at Week 52 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Time Frame: Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Number; unit: Percentage of participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 310 | 306 | 611
Percentage of participants | 70.6 | 72.5 | 78.6
Statistical Analysis 1: Comparison: 80 mg Ixekizumab Q4W vs 80 mg Ixekizumab Q2W; Test type: Superiority; p = 0.005, Regression, Logistic; Risk Difference (RD) = 7.9
Statistical Analysis 2: Comparison: 80 mg Ixekizumab Q4W vs 80 mg Ixekizumab Q4W/Q2W; Test type: Superiority; p = 0.522, Regression, Logistic; Risk Difference (RD) = 1.9

2. Primary Outcome: Percentage of Participants Achieving 75% Improvement in Psoriasis Area and Severity Index (PASI 75)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling, redness, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no Ps to 72 for the most severe disease. For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease). Participants who did not meet the clinical response criteria or had missing data at Week52 were considered non-responders for NRI analysis.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 310 | 306 | 611
Percentage of participants | 79 | 83.7 | 85.9
Statistical Analysis 1: Comparison: 80 mg Ixekizumab Q4W vs 80 mg Ixekizumab Q2W; Test type: Superiority; p = 0.006, Regression, Logistic; Risk Difference (RD) = 6.9
Statistical Analysis 2: Comparison: 80 mg Ixekizumab Q4W vs 80 mg Ixekizumab Q4W/Q2W; Test type: Superiority; p = 0.118, Regression, Logistic; Risk Difference (RD) = 4.6

3. Secondary Outcome: Percentage of Participants Achieving sPGA (0)
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's Ps was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline. Participants who did not meet the clinical response criteria or had missing data at Week 52 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 310 | 306 | 611
Percentage of participants | 44.8 | 48.7 | 60.1

4. Secondary Outcome: Percentage of Participants Achieving PASI 90
Description: PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling, redness, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no Ps to 72 for the most severe disease. For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 310 | 306 | 611
Percentage of participants | 65.2 | 73.9 | 79.5

5. Secondary Outcome: Percentage of Participants Achieving PASI 100
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling, redness, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no Ps to 72 for the most severe disease. For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no Ps) to 72 (the most severe disease).
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 310 | 306 | 611
Percentage of participants | 43.5 | 49.3 | 59.7

6. Secondary Outcome: Change From Baseline in PASI
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling, redness, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no Ps to 72 for the most severe disease.
  Least Squares mean (LSmean) was calculated using Mixed-Effects Model of Repeated Measures (MMRM) analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and had a baseline and post-baseline measurement for PASI. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 274 | 268 | 538
units on a scale | -18.34 (0.22) | -18.95 (0.22) | -19.41 (0.17)

7. Secondary Outcome: Percent Improvement in PASI
Description: as for outcome 6
Time Frame: Baseline, Week 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 274 | 268 | 538
Percent change | 91.09 (0.89) | 94.24 (0.90) | 96.25 (0.71)

8. Secondary Outcome: Mean Change From Baseline in Percent Body Surface Area (BSA) Involvement
Description: The percentage involvement of psoriasis on each participant's body surface area (BSA) was assessed by the investigator on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand including palm, fingers and thumb.
  LS mean was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned who had baseline and a post-baseline measurement for BSA affected by Psoriasis. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Percent Body Surface Affected
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 274 | 268 | 538
Percent Body Surface Affected | -23.93 (0.34) | -24.62 (0.34) | -25.01 (0.27)

9. Secondary Outcome: Mean Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score
Description: The NAPSI is a numeric, reproducible, objective tool for evaluation of fingernail (fn) Ps. This scale is used to evaluate the severity of fn bed Ps and fn matrix Ps by area of involvement in the fn unit. The fn is divided with imaginary horizontal and longitudinal lines into quadrants. Each fn is given a score for fn bed Ps (0 to 4) and fn matrix Ps (0 to 4) depending on presence (score of 1) or absence (score of 0) of any of the features of fn bed and fn matrix Ps in each quadrant. The NAPSI score of a fn is sum of scores in fn bed and fn matrix from each quadrant (maximum of 8). Each fn is evaluated, then the sum of all fn equals the total NAPSI score with a range from 0 to 80 (0 indicates no Ps, 80 indicates worst Ps). LS mean was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned who had baseline fingernail involvement and had a post-baseline measurement. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 156 | 148 | 314
units on a scale | -19.27 (0.81) | -19.87 (0.83) | -20.82 (0.62)

10. Secondary Outcome: Mean Change From Baseline in Psoriasis Scalp Severity Index (PSSI) Score
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90-100%) with a total score ranging from 0 (less severity) to 72 (more severity). LS mean change was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and had baseline scalp involvement and had a post-baseline measurement. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 252 | 245 | 477
units on a scale | -18.35 (0.31) | -18.73 (0.31) | -18.65 (0.24)

11. Secondary Outcome: Mean Change From Baseline in Palmoplantar PASI (PPASI)
Description: The Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 (no PPASI) to 72 (most severe PPASI). The PPASI was only assessed if participants have palmoplantar psoriasis at baseline. LS mean was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and had baseline palmoplantar Ps involvement and had post-baseline measurement. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 72 | 82 | 150
units on a scale | -9.55 (0.31) | -9.37 (0.30) | -9.00 (0.26)

12. Secondary Outcome: Percentage of Participants Achieving an Itch Numeric Rating Scale (Itch NRS) ≥4 Point Reduction From Baseline
Description: The Itch NRS is a participant-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours. Participants who did not meet the clinical response criteria or had missing data at Week 52 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and who had baseline Itch NRS score greater than or equal to (>=) 4. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups
Measure: Number; unit: Percentage of participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 254 | 260 | 505
Percentage of participants | 74.0 | 72.3 | 77.2

13. Secondary Outcome: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Total Score of 0 and 1 (DLQI [0,1])
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment). Participants who did not meet the clinical response criteria or had missing data at Week 52 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 310 | 306 | 611
Percentage of participants | 66.1 | 70.3 | 74.0

14. Secondary Outcome: Change From Baseline in DLQI Total Score
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment). LS mean change was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and who had baseline and post-baseline DLQI data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 273 | 265 | 538
units on a scale | -9.70 (0.21) | -9.97 (0.22) | -10.23 (0.17)

15. Secondary Outcome: Change From Baseline in Itch NRS Score
Description: The Itch NRS is a participant-administered single-item 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours. LS mean change from baseline in PSSI was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and who had baseline and post-baseline Itch NRS data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 274 | 268 | 537
units on a scale | -4.90 (0.13) | -5.15 (0.13) | -5.33 (0.10)

16. Secondary Outcome: Change From Baseline in Skin Pain Visual Analog Scale (VAS)
Description: The pain VAS is a participant-administered single-item scale designed to measure Skin pain from Psoriasis using a 0-100 millimeter (mm) horizontal VAS. Overall severity of participant's skin pain from Psoriasis is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no skin pain) to 100 mm (severe skin pain). LS mean was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and who had baseline and post-baseline skin pain VAS data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 271 | 262 | 532
mm | -35.50 (0.94) | -36.77 (0.96) | -38.07 (0.74)

17. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions 5 Level (EQ-5D-5L) VAS
Description: EQ-5D-5L is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of 2 components: a descriptive system of the respondent's health and a rating of his/her current health state using a 0 (no pain) to 100mm VAS (severe pain). LS mean was calculated using MMRM analysis including dosing regimen, country, baseline weight category, baseline value, visit, dosing regimen-by-visit, and baseline value-by-visit interactions as fixed factors, with variance-covariance structure set to unstructured.
Time Frame: Baseline, Week 52
Population: All randomized participants analyzed according to the treatment to which they were assigned and who had baseline and post baseline EQ-5D-5L VAS data. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 268 | 264 | 519
mm | 11.93 (0.94) | 12.47 (0.95) | 14.42 (0.74)

18. Secondary Outcome: Pharmacokinetics (PK): Trough Concentration at Steady State (Ctrough,ss) of Ixekizumab
Description: Trough concentrations at steady state of Ixekizumab were evaluated.
Time Frame: Predose, Week 4, 12, 24, 36 and 52 Post dose
Population: All randomized participants analyzed according to treatment to which they were assigned with evaluable PK samples that met the definition of being a trough concentration. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- 80 mg Ixekizumab Q4W Continuous: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q4W to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q4W/Q2W No Step: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as one SQ injection Q4W to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q4W/Q2W Step up: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as one SQ injection Q4W with step-up dosing to Q2W as needed (Q4W/Q2W step-up) to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q2W Continuous: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q2W to week 52. Placebo administered SQ, Q2W to maintain blind.
Arm/Group | 80 mg Ixekizumab Q4W Continuous | 80 mg Ixekizumab Q4W/Q2W No Step | 80 mg Ixekizumab Q4W/Q2W Step up | 80 mg Ixekizumab Q2W Continuous
Number analyzed (Participants) | 304 | 232 | 73 | 602
microgram per milliliter (µg/mL)
  Week 4 | 3.55 (76) | 4.03 (72) | 2.78 (67) | 7.87 (63)
  Week 12 | 2.72 (72) | 2.81 (80) | 1.95 (70) | 8.23 (56)
  Week 24 | 2.65 (73) | 2.71 (85) | 3.48 (78) | 7.89 (66)
  Week 36 | 2.83 (74) | 2.88 (73) | 5.76 (67) | 7.73 (76)
  Week 52 | 2.43 (79) | 2.77 (73) | 5.73 (68) | 6.96 (87)

19. Secondary Outcome: Number of Participants With Anti-Ixekizumab Antibodies
Description: Number of participants with treatment-emergent positive anti-ixekizumab antibodies was summarized by treatment group.
Time Frame: Baseline through Week 52
Population: All randomized participants who received at least 1 dose of Ixekizumab and had evaluable anti-ixekizumab antibody measurement. As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Number; unit: participants
Arm/Group | 80 mg Ixekizumab Q4W | 80 mg Ixekizumab Q4W/Q2W | 80 mg Ixekizumab Q2W
Number analyzed (Participants) | 307 | 305 | 606
participants | 71 | 64 | 84

ADVERSE EVENTS:
Time Frame: Up to 19 months
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Ixekizumab 80 mg Q4W - Treatment Period; 80 mg Ixekizumab Q4W - Treatment Period ME2 Cohort: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q4W to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q4W/Q2W - Treatment Period; 80 mg Ixekizumab Q4W/Q2W - Treatment Period ME2 Cohort: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as one SQ injection Q4W with step-up dosing to Q2W as needed (Q4W/Q2W step-up) to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q2W - Treatment Period; 80 mg Ixekizumab Q2W - Treatment Period ME2 Cohort: 160 mg ixekizumab given as 2 SQ injections at baseline and then 80 mg ixekizumab given as 1 SQ injection Q2W to week 52. Placebo administered SQ, Q2W to maintain blind.
- 80 mg Ixekizumab Q4W - Post-Treatment Period; 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period; 80 mg Ixekizumab Q2W - Post-Treatment Period; 80 mg Ixekizumab Q4W - Post-Treatment Period ME2 Cohort; 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period ME2 Cohort; 80 mg Ixekizumab Q2W - Post-Treatment Period ME2 Cohort: Participants didn't receive any intervention.
Arm/Group | Ixekizumab 80 mg Q4W - Treatment Period | 80 mg Ixekizumab Q4W/Q2W - Treatment Period | 80 mg Ixekizumab Q2W - Treatment Period | 80 mg Ixekizumab Q4W - Post-Treatment Period | 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period | 80 mg Ixekizumab Q2W - Post-Treatment Period | 80 mg Ixekizumab Q4W - Treatment Period ME2 Cohort | 80 mg Ixekizumab Q4W/Q2W - Treatment Period ME2 Cohort | 80 mg Ixekizumab Q2W - Treatment Period ME2 Cohort | 80 mg Ixekizumab Q4W - Post-Treatment Period ME2 Cohort | 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period ME2 Cohort | 80 mg Ixekizumab Q2W - Post-Treatment Period ME2 Cohort
All-Cause Mortality (participants affected / at risk) | 0/310 | 0/306 | 0/609 | 0/285 | 0/283 | 0/559 | 0/9 | 0/5 | 0/16 | 0/9 | 0/4 | 0/15
Serious Adverse Events (participants affected / at risk) | 16/310 | 16/306 | 32/609 | 1/285 | 2/283 | 7/559 | 0/9 | 1/5 | 0/16 | 0/9 | 0/4 | 0/15
Other Adverse Events (participants affected / at risk) | 157/310 | 136/306 | 285/609 | 16/285 | 20/283 | 40/559 | 6/9 | 4/5 | 11/16 | 2/9 | 0/4 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab 80 mg Q4W - Treatment Period (N=310) | 80 mg Ixekizumab Q4W/Q2W - Treatment Period (N=306) | 80 mg Ixekizumab Q2W - Treatment Period (N=609) | 80 mg Ixekizumab Q4W - Post-Treatment Period (N=285) | 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period (N=283) | 80 mg Ixekizumab Q2W - Post-Treatment Period (N=559) | 80 mg Ixekizumab Q4W - Treatment Period ME2 Cohort (N=9) | 80 mg Ixekizumab Q4W/Q2W - Treatment Period ME2 Cohort (N=5) | 80 mg Ixekizumab Q2W - Treatment Period ME2 Cohort (N=16) | 80 mg Ixekizumab Q4W - Post-Treatment Period ME2 Cohort (N=9) | 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period ME2 Cohort (N=4) | 80 mg Ixekizumab Q2W - Post-Treatment Period ME2 Cohort (N=15)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular stent restenosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cartilage hypertrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basilar migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/111 (0) | 0/107 (0) | 0/199 (0) | 0/98 (0) | 0/98 (0) | 1/184 (1) | 0/2 (0) | 0/0 (0) | 0/4 (0) | 0/2 (0) | 0/0 (0) | 0/4 (0)
Tubal rupture (Pregnancy, puerperium and perinatal conditions) | 0/111 (0) | 0/107 (0) | 0/199 (0) | 0/98 (0) | 0/98 (0) | 1/184 (1) | 0/2 (0) | 0/0 (0) | 0/4 (0) | 0/2 (0) | 0/0 (0) | 0/4 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/199 (1) | 0/199 (0) | 0/410 (0) | 0/187 (0) | 0/185 (0) | 0/375 (0) | 0/7 (0) | 0 (0) | 0/12 (0) | 0/7 (0) | 0 (0) | 0/11 (0)
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab 80 mg Q4W - Treatment Period (N=310) | 80 mg Ixekizumab Q4W/Q2W - Treatment Period (N=306) | 80 mg Ixekizumab Q2W - Treatment Period (N=609) | 80 mg Ixekizumab Q4W - Post-Treatment Period (N=285) | 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period (N=283) | 80 mg Ixekizumab Q2W - Post-Treatment Period (N=559) | 80 mg Ixekizumab Q4W - Treatment Period ME2 Cohort (N=9) | 80 mg Ixekizumab Q4W/Q2W - Treatment Period ME2 Cohort (N=5) | 80 mg Ixekizumab Q2W - Treatment Period ME2 Cohort (N=16) | 80 mg Ixekizumab Q4W - Post-Treatment Period ME2 Cohort (N=9) | 80 mg Ixekizumab Q4W/Q2W - Post-Treatment Period ME2 Cohort (N=4) | 80 mg Ixekizumab Q2W - Post-Treatment Period ME2 Cohort (N=15)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 4 (14) | 3 (4) | 18 (49) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (24) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (24) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (4) | 6 (7) | 8 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (4) | 0 (0) | 4 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 18 (68) | 5 (15) | 49 (256) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 2 (11) | 0 (0) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 3 (3) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 4 (7) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 6 (6) | 9 (10) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 3 (4) | 3 (4) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 6 (6) | 4 (4) | 8 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 46 (60) | 39 (56) | 69 (93) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 16 (21) | 4 (4) | 15 (20) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/111 (0) | 1/107 (1) | 0/199 (0) | 0/98 (0) | 0/98 (0) | 0/184 (0) | 0/2 (0) | 0/0 (0) | 1/4 (1) | 0/2 (0) | 0/0 (0) | 0/4 (0)
Viral upper respiratory tract infection (Infections and infestations) | 41 (49) | 53 (69) | 73 (89) | 6 (7) | 0 (0) | 9 (9) | 1 (1) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (5) | 25 (29) | 2 (3) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 14 (16) | 16 (18) | 29 (34) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 2 (3) | 23 (25) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 17 (17) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 6 (8) | 5 (6) | 11 (12) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 3 (3) | 3 (4) | 5 (5) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days